CLINICAL TRIAL: NCT05858294
Title: The Safety, Acceptability and Efficacy of Alena, a Modularized CBT-based Mobile App Intervention for Social Anxiety: a Randomised Controlled Trial
Brief Title: The Safety, Acceptability and Efficacy of Alena
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aya Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Alena CBT RCT 2022
Record Dates: First submitted 2023-04-21; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Social Anxiety; Social Anxiety Disorder; Social Anxiety Disorder (Social Phobia)
Keywords: RCT; CBT
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy program (Experimental): Access to the "Alena" CBT-based therapy programme for 4 weeks. Each of the four therapy modules gradually became available on a weekly basis until all four were available in the final intervention week. Participants were instructed to complete one module per week. Each therapy module consisted of psychoeducational content, guided psychological reflection and perspective-taking exercises, and, where appropriate, skills training exercises such as attention training, public speaking, and exposure experiments to be completed in real life.
  Interventions: Behavioral: Cognitive Behavioral Therapy programme
- Waitlist control (No Intervention): Waitlist control. Participants in this arm were given access to the CBT content at the end of the 4-week trial period.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy programme — This mobile application comprised CBT-based therapy for social anxiety based on the Clark and Wells model
  Arms: Cognitive Behavioral Therapy program

SUMMARY:
The present study is a randomised controlled trial that seeks to investigate the safety, acceptability and efficacy and safety of the Alena CBT programme as a treatment for social anxiety disorder.

DETAILED DESCRIPTION:
This is a 6-week web-based parallel-group unblinded randomised controlled trial with a 4-week intervention period and a 2-week follow-up post intervention. Participants are randomly allocated to receive access to the Alena CBT programme or to a wait list control group, in a 1:1 ratio. The programme consists of CBT-based therapy for social anxiety based on the Clark and Wells model.

ELIGIBILITY:
Inclusion Criteria:

* female
* aged between 18 and 35 years old (inclusive)
* located in the UK
* fluent in English
* comfortable taking part in a study that included deception (due to the nature of the cognitive assessments)
* had an iPhone and daily access to an internet connection
* scored over 30 on the Social Phobia Inventory (SPIN; indicating at least moderate social anxiety).

Exclusion Criteria:

* currently undergoing any mental health therapy
* changed the usual mental health medication or dosage within the past eight weeks
* scored eight or above on the Alcohol Use Disorders Identification Test for consumption (AUDIT-C; indicating higher risk of alcohol dependence)
* scored two or above on the adapted drug questions (indicating higher risk of drug dependence)
* had previously participated in scientific studies or user research undertaken by Alena

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Questionnaires assessing negative effects from using the app and adverse health events | Week 4 (primary endpoint)
  The Intervention group was asked "Have you experienced any negative effects from using the Alena app? This could be a physical or emotional effect that you believe you have experienced as a result of using the app and/or engaging in the app therapy." Both groups were asked: "Have you experienced any new, serious negative health effects in the past week? This includes having to see your GP for a new reason, going to hospital, or being otherwise very unwell in terms of your physical or mental health." If participants responded positively to either question, they were prompted for additional details and to rate the severity of the experience.
Questionnaires assessing negative effects from using the app and adverse health events | Week 6 (2-week follow-up post-intervention)
  The Intervention group was asked "Have you experienced any negative effects from using the Alena app? This could be a physical or emotional effect that you believe you have experienced as a result of using the app and/or engaging in the app therapy." Both groups were asked: "Have you experienced any new, serious negative health effects in the past week? This includes having to see your GP for a new reason, going to hospital, or being otherwise very unwell in terms of your physical or mental health." If participants responded positively to either question, they were prompted for additional details and to rate the severity of the experience.
Questionnaire assessing satisfaction, helpfulness and ease of use | Week 4 (primary endpoint)
  Participants were asked how satisfied they were with the app overall (Likert rating scale from very dissatisfied to very satisfied); how helpful they found the app (Likert ratings from very unhelpful to very helpful); how likely they would be to recommend the app (Likert ratings from very unlikely to very likely); how easy they found using the app (Likert ratings from very difficult to very easy); whether they got to the end of the weekly exercise (yes/no), and what got in the way of completing the exercises, with options provided.
Questionnaire assessing satisfaction, helpfulness and ease of use | Week 6 (2-week follow-up post-intervention)
  Participants were asked how satisfied they were with the app overall (Likert rating scale from very dissatisfied to very satisfied); how helpful they found the app (Likert ratings from very unhelpful to very helpful); how likely they would be to recommend the app (Likert ratings from very unlikely to very likely); how easy they found using the app (Likert ratings from very difficult to very easy); whether they got to the end of the weekly exercise (yes/no), and what got in the way of completing the exercises, with options provided.

SECONDARY OUTCOMES:
Social phobia inventory (SPIN) | Week 4 (primary endpoint)
  The SPIN was designed to assess the full spectrum of symptoms that characterise social anxiety, including fear, avoidance and physiological components. Total score ranging from 0 to 68, with higher scores indicating a worse outcome.
Social phobia inventory (SPIN) | Week 6 (2-week follow-up post-intervention)
  The SPIN was designed to assess the full spectrum of symptoms that characterise social anxiety, including fear, avoidance and physiological components. Total score ranging from 0 to 68, with higher scores indicating a worse outcome.
Work and Social Adjustment Scale (WSAS) | Week 4 (primary endpoint)
  The WSAS measures the extent to which the respondent's problem impairs their ability to carry out day-to-day activities, such as work, home management and social leisure activities. Total score ranging from 0 to 40, with higher scores indicating higher impairment
Work and Social Adjustment Scale (WSAS) | Week 6 (2-week follow-up post-intervention)
  The WSAS measures the extent to which the respondent's problem impairs their ability to carry out day-to-day activities, such as work, home management and social leisure activities. Total score ranging from 0 to 40, with higher scores indicating higher impairment

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Ahmadi, PhD, Principal Investigator — Aya Technologies Limited
Locations (1):
- Aya Technologies Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Connor KM, Davidson JR, Churchill LE, Sherwood A, Foa E, Weisler RH. Psychometric properties of the Social Phobia Inventory (SPIN). New self-rating scale. Br J Psychiatry. 2000 Apr;176:379-86. doi: 10.1192/bjp.176.4.379. PMID 10827888
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Derived] Garvert MM, McFadyen J, Linke S, McCloud T, Meyer SS, Sobanska S, Sharp PB, Long A, Huys QJM, Ahmadi M. Safety and Efficacy of Modular Digital Psychotherapy for Social Anxiety: Randomized Controlled Trial. J Med Internet Res. 2025 Apr 10;27:e64138. doi: 10.2196/64138. PMID 40208666